CLINICAL TRIAL: NCT01849978
Title: Enhancing Exercise in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Pro00044422
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; survivor; exercise; physical activity; strenuous exercise; moderate exercise; enjoyable exercise; enjoy exercise; breast cancer survivor
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Active Comparator): Participants in this arm will receive the newsletter about their reported minutes of physical activity and the benefits of physical activity specific to breast cancer survivors, and the brochure "Changing your habits," developed by the NIH.
  Interventions: Behavioral: Newsletter about physical activity and breast cancer survivors; Behavioral: Changing your habits brochure
- Habit Formation Arm (Active Comparator): Participants in this arm will receive all of the intervention materials.
  Interventions: Behavioral: Newsletter about physical activity and breast cancer survivors; Behavioral: Changing your habits brochure; Behavioral: Tips for making exercise enjoyable and personally-valued; Behavioral: Testimonials from breast cancer survivors

INTERVENTIONS:
Behavioral: Newsletter about physical activity and breast cancer survivors — Both groups will receive a newsletter that covers: 1) the recommendation to pursue at least 150 mins/week of moderate to strenuous intensity PA, 2) the benefits of PA specific to breast cancer survivors (e.g., reducing in death and breast cancer recurrence), and 3) their total minutes of moderate to strenuous intensity PA and how this compares to the recommendation.
Behavioral: Changing your habits brochure — Both groups will receive the brochure titled "Changing Your Habits: Steps to Better Health", developed by the NIH, that describes, based a person's stage of change, the benefits of PA, how to overcome common barriers to PA, and if ready, how to plan for PA.
Behavioral: Tips for making exercise enjoyable and personally-valued — Participants will get a list of potentially enjoyable activities and a space to list other activities after they consider aspects that can make events fun/interesting.13 Aspects to consider include: location (indoors vs. outdoors, the latter which may appeal to some), hobbies that can involve PA (e.g., sports, dancing), whether the activity is made more enjoyable by having it performed by oneself or with others (e.g., team activities vs. individual activities); what valued outcomes may be achieved (e.g., sense of competence, pride, better health, body image), accompanying activities that are pleasant (e.g., listening to music), etc.
  Arms: Habit Formation Arm
Behavioral: Testimonials from breast cancer survivors — Participants will get two to three testimonials of actual breast cancer survivors. These testimonials will include story-like details of what these survivors find enjoyable about exercising and what they have done to make exercise enjoyable.
  Arms: Habit Formation Arm

SUMMARY:
This study will examine whether or not providing early stage breast cancer survivors with tips on making exercise more enjoyable promotes greater levels of moderate to strenuous exercise.

ELIGIBILITY:
Inclusion Criteria:

* no health restrictions on performing moderate to strenuous physical activity
* must be 18 years or older and able to give legal consent

Exclusion Criteria:

* may not be participating in another research study regarding exercise
* restrictions on performing physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
change in number of minutes of moderate to strenuous physical activity | baseline, 1 month and 3 months
  participants will self-report minutes of physical activity at baseline, 1 month, and 3 months after receiving intervention materials.

SECONDARY OUTCOMES:
changes in joy and satisfaction with physical activity | baseline, 1 month, and 3 months
  participants will self-report via questionnaire their joy and satisfaction with their average physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Lipkus, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States